CLINICAL TRIAL: NCT03145129
Title: Positive Airway Pressure and Intraocular Relationship: Study 2- The Impact of CPAP on Nocturnal IOP.
Brief Title: PAIR Study-PAP And IOP Relationship: Study 2
Acronym: PAIR2
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Hinchingbrooke Healthcare NHS Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: P02145
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnoea; Primary Open-angle Glaucoma
Keywords: Intraocular pressure; IOP; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glaucoma, Open-Angle | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAG group: Patients diagnosed with POAG and OSA who require treatment with CPAP
  Interventions: Device: Continuous Positive Airway Pressure
- Control group: Patients with OSA and without POAG who require treatment with CPAP
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure

SUMMARY:
Some people with Primary Open-angle Glaucoma (POAG) also suffer from Obstructive Sleep Apnoea (OSA), a common sleep disorder which is known to affect heart and blood vessels, and may contribute to glaucoma progression. Obstructive Sleep Apnoea is treated with Continuous Positive Airway Pressure (CPAP); however using this type of breathing support may raise intraocular pressure (IOP). The evidence for this is limited and the potential mechanisms involved are poorly understood.

In this study we will determine whether CPAP applied at night changes IOP and ocular perfusion pressure (OPP). We will also assess its possible impact on ocular microvasculature. Two groups of patients will be included: those with POAG and OSA, and those with OSA without glaucoma. They will attend for two overnight assessments: the first before starting CPAP and the second 4-6 weeks into the treatment. Repeated measurements of IOP at night will be performed and participants will continue self-measuring IOP at home in the day. An Ocular Coherence Tomography Angiography (OCT Angiography) of the optic disc and the surrounding retina will be performed at baseline and after a few weeks of CPAP treatment.

DETAILED DESCRIPTION:
People with OAG and concomitant OSA associated with the relevant symptoms, particularly daytime sleepiness, currently receive standard treatment with CPAP. However, the impact of CPAP on their glaucoma is unknown. There are concerns that CPAP increases IOP, currently the only modifiable factor in glaucoma, though the evidence for this is limited.

Understanding the influence of CPAP on IOP is important as it may inform the management of people with OSA and concomitant glaucoma. If CPAP is shown to raise IOP or alter OPP to levels that pose clinical risk it will be necessary to assess available alternative treatment options for OSA. If, however, CPAP does not alter these parameters, there would be a rationale for assessing long-term effects of CPAP, most probably in the form of a randomised interventional trial, informed by the findings of this research.

This is a prospective controlled study which will examine the impact of CPAP on nocturnal IOP and OPP in people with OSA with and without POAG. In addition, we will assess ocular microvasculature before and a few weeks into CPAP treatment.

Objectives:

Primary: to determine if IOP increases at night following treatment with CPAP in people with OSA with and without POAG.

Main Secondary:(i) to investigate whether diurnal IOP raises after CPAP treatment; (ii) to investigate whether CPAP alters peri-papillary and macular microcirculation measured with OCT Angiography.

Participants: People with newly diagnosed OSA who require treatment with CPAP will be invited. We will recruit participants with POAG and people without glaucoma (control subjects). All participant will undergo a detailed ocular assessment including: visual acuity, IOP measurement, OCT and visual field test.

Sample Size: 30 participants: 15 per group.

Study Visits:

Visit 0: Baseline ocular examination to confirm or exclude glaucoma will be undertaken during this visit unless a participant already had this examination within the last 6 months.

Visit 1: Participants will attend the sleep centre (Respiratory Support and Sleep Centre-RSSC, Papworth Hospital) where they will be admitted to a separate ward. Consented participants will undergo the following:

Baseline assessment: A brief medical history, spirometry and anthropomorphic measurements.

Repeated measurements: IOP will be measured in each eye using a rebound tonometer (Icare Pro, Finland Oy). Blood pressure and ocular perfusion pressure will be checked simultaneously.

Participants will be advised to sleep at their habitual hours. Sleep onset and duration will be recorded. All the above measurements will be repeated every 2 hours starting from 10pm and finishing at 8am. In the morning OCT Angiographic will be performed.

Participants will then self-measure IOP at home using a rebound tonometer (Icare Home, Finland Oy). The measurements will be performed in the daytime every 2 hours before they start CPAP and 4-6 weeks into the treatment.

Visit 2: Participants will return for the second overnight assessment 4-6weeks after initiation of CPAP treatment.

CPAP usage data will be downloaded. All the measurements following the same procedure as for Visit 1 will be repeated this time with participants using CPAP. OCT Angiographic will be performed immediately after removing CPAP in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, untreated OSA with indications for CPAP
* Age >40 years
* Able to give informed consent and attend for the study visits.

Exclusion Criteria:

* Known or suspected pregnancy
* Any contraindications to rebound tonometry, including: corneal scarring, microphtalmos, buphthalmos, nystagmus, keratoconus, abnormal central corneal thickness, corneal ectasia, , active corneal infection, , and corneal dystrophies
* Eye diseases known to affect IOP, including: treated wet age related macular degeneration (ARMD), central retinal vein occlusion (CRVO), branch retinal vein occlusion (BRVO), uveitis and diabetic retinopathy.
* Indications to start CPAP treatment urgently unless the study visits can be organised in a way there is no delay in treatment initiation.
* Irregular sleep pattern
* Insomnia
* Acute infectious diseases
* Inability to undergo screening ophthalmic examination

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are two recruitment sources:
  i. Eligible participants who have completed the POSAG trial (NCT02713152) and were diagnosed with OSA for which CPAP treatment was recommended.
  ii. Patients who attend Sleep Disturbance Clinic (SDC) at Papworth.
  We aim to recruit 15 participants with OSA and POAG (Glaucoma group) and 15 participants with OSA and no Glaucoma (Control group). Patients with OSA and POAG will be recruited first and control participants matched for OSA severity subsequently. Matching will be performed according to 3 OSA categories: mild (AHI:5-15), moderate (AHI:15-30), severe (AHI>30)).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | On completion of study visit 2: 6 weeks
  Difference between baseline IOP at night and nocturnal IOP on CPAP

SECONDARY OUTCOMES:
Diurnal IOP change | On completion of study visit 2: 6 weeks
  A difference in diurnal IOP self-measured at home at baseline and during CPAP treatment.
Differences in change in IOP between the study group | On completion of study visit 2: 6 weeks
  Differences in IOP change (ΔIOP; IOPCPAP -IOPbaseline) between the groups
Relationship between change in IOP on CPAP with OSA severity | On completion of study visit 2: 6 weeks
  Correlation between IOP change (ΔIOP) and AHI (Apnoea-Hypopnoea Index)
Relationship between change in IOP on CPAP with POAG severity | On completion of study visit 2: 6 weeks
  Correlation between IOP change (ΔIOP) and VFI (Visual Field Index)
Ocular Perfusion Pressure (OPP) | On completion of study visit 2: 6 weeks
  Difference between baseline OPP at night and nocturnal OPP on CPAP in each group
Optic disc vessel density | On completion of study visit 2: 6 weeks
  Optic disc vessel density at baseline and after 4-6 weeks of CPAP treatment
Peripapillary vessel density | On completion of study visit 2: 6 weeks
  Peripapillary vessel density at baseline and after 4-6 weeks of CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Wozniak, MBBS, MRCP, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No